CLINICAL TRIAL: NCT02922504
Title: Impact of Music Intervention on Pain Control In First Trimester Surgical Abortion Under Local Anesthesia
Acronym: AlgoMusic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 49RC16_0073
Record Dates: First submitted 2016-09-27; First posted 2016-10-04 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: First Trimester Abortion; Surgical Abortion; Music Intervention; Local Anesthesia; Pain
Keywords: First trimester abortion; Surgical abortion; Music intervention; Local anesthesia; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Music intervention group (Experimental): For the patients in the Music intervention group, a adjuvant treament by a music intervention will be use before the procedure
  Interventions: Behavioral: Music intervention group
- Controlled group (Active Comparator): For the patients in the " controlled " group, the use of analgesic will be use if needed during the procedure
  Interventions: Behavioral: Controlled group

INTERVENTIONS:
Behavioral: Music intervention group
  Arms: Music intervention group
Behavioral: Controlled group
  Arms: Controlled group

SUMMARY:
A surgical abortion under local anesthesia is potentially painful. A protocol using analgetic is systematically used. Also the protocol is relevant , the question of taking care of the pain in a safe manner remains.

The use of Music during surgery can have a real effect on pain and anxiety. This study has for goal to evalued the use of music on pain as adjuvant treatement instead of a standard care for an abortion.

DETAILED DESCRIPTION:
A surgical abortion under local anesthesiac is potentially painful. A protocol using analgetic is systematically used. Also the protocol is relevant, the question of taking care of the pain in a safe manner remains.

The use of Music during surgery can have a real effect on pain and anxiety. This study has for goal to evalued the use of music on pain as adjuvant treatment instead of a standard care for an abortion.

The number of patients needed is estimate to be eighty patients per group.

The result of the study could allow :

* Showing the effectiveness of music intervention before operative abortion as adjuvant treatment on the pain, anxiety and nausea during a surgical abortion by suction aspiration under local anesthesia.
* Improving the experience of an abortion and the satisfaction of the patients as well as lowering the use of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Every patients must have more than 18 years old
* Hospitalised at the Angers Hospital for a surgical abortion under local anesthesia.
* Affiliated or be part of the french Sécurité Sociale ( health service )
* To have signed a consent form

Exclusion Criteria:

* Patients not speaking french
* People who should not use music intervention ( Total or partial hearing difficulties)
* No consent given
* Adults protected by the law
* Not being part of another medical study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-10; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
the effectiveness on the pain of music therapy by the pain evaluation with visual numeric scale | during one day
  evaluation is maide five times